CLINICAL TRIAL: NCT04548908
Title: Prevalence Of COVID-19 Among Health-workers in a French General Hospital
Acronym: POCAH-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Sud Essonne (Other)
Responsible Party: Sponsor
Other Study IDs: POCAH-COVID19
Record Dates: First submitted 2020-09-07; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: health-workers; COVID19; hospital; SARS-CoV-2; prevalence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Serelogy testing, RT PCR — Serology testing for all the participants and RT PCR for participants with symptoms

SUMMARY:
The aim of this study is to evaluate the prevalence of COVID-19 among the workers of our hospital and the factors that are likely to influence this prevalence. It must be underlined that our hospital is settled in two towns and both hospital sites had different missions regarding the admissions of COVID-19-infected patients.

DETAILED DESCRIPTION:
Since December 2019, the COVID-19 pandemic has widespread from China and put under strong tension the health organizations throughout the world, especially since march 2020 in France.

As a consequence, the French hospitals had to cope with a massive amount of COVID-19 infected patients and, thus, their organisations had to evolve in order to be able to admit more patients in their critical care units.

First studies reported an important level of inter-human contagiousness of the SARS-CoV-2 virus with an "R0" (basic reproduction number) superior to 3, which could lead to a massive contamination of healthcare workers since they are directly in charge of infected patients.

Other studies suggested that the healthcare workers are more likely to be contaminated by the COVID-19 than the rest of the population, which pushed governments and hospital managers to put in place individual and collective measures of protection in order to avoid nosocomial transmissions and also to preserve the health of the hospital staffs in a context of high tension on the hospital work force.

There are today few data about the contamination level among the healthcare workers of general hospitals in France and about the severity of these contaminations. A national study is being conducted but on a macroscopic regional scale. In addition to that, the proportion of asymptomatic SARS-CoV-2 contaminated healthcare workers is not known as well as the origin (hospital or community) of the contaminations.

In June 2020, the French Health Ministry decided to launch a collection of epidemiological data in the French hospitals based on serologic tests. Thanks to this action and with the results of all the RT PCR tests systematically conducted since the beginning of the pandemic when a healthcare worker had COVID-19-like symptoms, the Centre Hospitalier Sud Essonne has decided to conduct an observational study.

The aim of this study is to evaluate the prevalence of COVID-19 among the workers of our hospital and the factors that are likely to influence this prevalence. It must be underlined that our hospital is settled in two towns and both hospital sites had different missions regarding the admissions of COVID-19-infected patients.

ELIGIBILITY:
Inclusion criteria:

* hospital staff working at the Centre Hospitalier Sud Essonne,
* employed by the Centre Hospitalier Sud Essonne between March, 5th, 2020, and August, 31rst, 2020,
* with the result of an RT PCR test or a serologic test,
* this (these) result(s) must have been/be communicated to the occupational health service of the hospital.

Exclusion criteria:

* interim workers,
* workers in holidays during the entire period of inclusion above,
* opposition to participate in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult healthcare workers who are not opposed to participate to the research
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
General prevalence of COVID-19 | Through study completion, an average of 9 months
  measures the prevalence of COVID-19 among the healthcare workers of the Centre Hospitalier Sud Essonne, defined as the hospital employees with positive serologic or RT-PCR tests.
  It must be underlined that the notion of "health workers" include the entire hospital staff ie doctors, nurses, administrative employees,...

SECONDARY OUTCOMES:
Number of asymptomatic healthcare workers | Through study completion, an average of 9 months
  * no RT PCR or negative RT PCR and positive serologic test,
  * positive RT PCR and no symptoms,
Number of symptomatic healthcare workers | Through study completion, an average of 9 months
  Positive RT-PCR test or serologic test with symptoms.
Number of healthcare workers with a severe form of COVID-19 which led to an hospitalization | Through study completion, an average of 9 months
  Positive serologic or RTC-PCR test and hospitalization
Number of healthcare workers infected with COVID-19 and hospitalized in a critical care unit | Through study completion, an average of 9 months
  Positive serologic or RTC-PCR test and hospitalization in a critical care unit
Influencing factors of the prevalence of the COVID-19 among healthcare workers | Through study completion, an average of 9 months
  * age,
  * gender,
  * job,
  * duration of employment in the hospital,
  * hospital site of affectation,
  * unit of affectation.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine LEMAIRE-BRUNEL, Principal Investigator — Centre Hospitalier Sud Essonne
Locations (1):
- Centre Hospitalier Sud Essonne, Étampes, France